CLINICAL TRIAL: NCT04072926
Title: Clinical Research of the Effects of Photodynamic Therapy and Bioceramic Filling of Root Canals on the Healing of Periapical Lesions and the Occurence of Postoperative Pain After Endodontic Retreatment
Brief Title: Effects of PDT and Bioceramic Filling on Periapical Healing and Postoperative Pain After Endodontic Retreatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical Innovation Center Wroclaw (Other)
Collaborators: University of Zagreb (Other)
Responsible Party: Principal Investigator, BORIS PAZIN, DDM, SPECIALIST IN ENDODONTICS AND RESTORATIVE DENTISTRY, Medical Innovation Center Wroclaw
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 021/002-19-208
Record Dates: First submitted 2019-08-27; First posted 2019-08-28 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Apical Periodontitis
Keywords: Biomaterials; irrigation protocol; pariapical healing
MeSH Terms: conditions — Periapical Periodontitis | interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Each of the two main groups are divided to two subgroups.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PDT+/BIOROOT (Experimental): Photodynamic therapy will bi conducted with diode laser (660nm, 100mW, 60 seconds) with toluidine at the end of chemomechanical preparation. Final root canal filling will be with BioRoot in combination with guttapercha points.
  Interventions: Drug: BioRoot
- PUI/BIOROOT (Experimental): This arm will only get PUI (passive ultrasound irrigation) with 2,5ml of 2,5% sodium hypochlorite, then 2ml of 15% EDTA which will be activated for 60seconds (EndoUltra MicroMega, France) and finally 2,5ml of 2,5% of sodium hypochlorite will be also activated for 30 seconds. Root canal filling in combination with BioRoot and guttapercha points.
  Interventions: Drug: BioRoot
- PDT+/AH+ (Active Comparator): Photodynamic therapy will bi conducted with diode laser (660nm, 100mW, 60 seconds) with toluidine at the end of chemomechanical preparation. Final root canal filling will be with AH+ epoxy based cement in combination with guttapercha points.
  Interventions: Drug: BioRoot
- PUI/AH+ (Active Comparator): This arm will only get PUI (passive ultrasound irrigation) in combination with AH+ epoxy based cement and guttapercha points.
  Interventions: Drug: BioRoot

INTERVENTIONS:
Drug: BioRoot — Influence of biomaterial BioRoot on periapical healing
  Other Names: Photodynamic therapy

SUMMARY:
The purpose is to investigate influence of bioceramic filling of the root canal and photodynamic therapy on periapical healing and development of postoperative pain after endodontic retreatment. Patients are divided into two main groups and each of the group is divided into two subgroups. Main groups are patients receiving photodynamic therapy and patients receiving passive ultrasonic irrigation. Each of the main group is divided by the root canal filling material on the AH+ group and BioRoot group.

DETAILED DESCRIPTION:
Clinical trial will be conducted in Dental clinic Zagreb. Patients will be chosen for this randomized prospective trials from the everyday patients referred by general dentist for endodontic retreatment. In the research will be included only patients with symptoms of chronic apical periodontitis and previous endodontic treatment. It includes teeth sensitive to palpation, percussion or visible sinus tract or swelling and asymptomatic inadequate endodontic filling. Patients that are immunocompromised, pregnant women, teeth with pocket depth bigger then 3mm, teeth with signs of vertical root fracture, teeth that are impossible to restore are excluded from research.

Every patient will be assigned to one group and one subgroup using "wheeldecide" programme. Patients will not be aware what group or subgroup they are assigned. endodontic retreatment will be conducted by one specialist in endodontics. Therapy is single visit retreatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of periapical disease after endodontic treatment,
* teeth sensitive to percussion and palpation,
* teeth with present sinus tract and
* asymptomatic teeth with radiologically inadequate root canal filling.

Exclusion Criteria:

* Immunocompromised patients,
* pregnancy,
* teeth with signs of vertical root fracture,
* teeth that can't be restored,
* antibiotic usage within last month,
* teeth with acute apical abscess

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in volume of periapical lesion | 1 year
  Volumetric change of size of periapical lesion depending of the root canal filling material and the use of photodynamic therapy at the end of chemomechanical preparation.
Level of postoperative pain after endodontic treatment | 7 days day after day monitoring of the level of pain.
  After endodontic treatment receives questionaire with day - by - day monitoring of the level of pain on the scale from 0 (no pain) to 10 (sever pain)

CONTACTS AND LOCATIONS:
Overall Officials: BORIS PAZIN, DDM, Principal Investigator — DENTAL CLINIC ZAGREB
Locations (1):
- Dental Clinic Zagreb, Zagreb, Croatia

REFERENCES:
- [Derived] Pazin B, Lauc T, Petricevic GK, Gabric D, Bago I. Periapical Lesion Healing After Retreatment and Root Canal Filling with a Bioceramic-Based Sealer: A Randomized Clinical Study with 1-Year Follow-Up. J Clin Med. 2025 Nov 21;14(23):8267. doi: 10.3390/jcm14238267. PMID 41375569